CLINICAL TRIAL: NCT07042074
Title: Use of a Spatial Computing Device and Augmented Reality and Virtual Reality for Exposure Therapy for Needle and Blood-Injection-Injury Phobia
Brief Title: Use of Augmented Reality and Virtual Reality During Cognitive Behavioral Therapy for Needle Phobia
Acronym: SNAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 77696
Record Dates: First submitted 2024-11-05; First posted 2025-06-27 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Needle Phobia; Virtual Reality; Cognitive Behavior Treatment
MeSH Terms: interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Behavioral Therapy (CBT) + Extended reality exposure therapy (XRET) (Experimental)
  Interventions: Behavioral: Mixed reality (XR) Exposure Therapy

INTERVENTIONS:
Behavioral: Mixed reality (XR) Exposure Therapy — Participants will engage in a minimum 8-session intervention combining Cognitive Behavioral Therapy (CBT) and Extended Reality Therapy (XRET) to address needle phobia and blood-injection-injury (BII) phobia. The intervention begins with an initial intake session where the APA-SMS screener results are reviewed. Participants will then undergo VR exposure, with mixed exposure to sham needles in the latter exposure session. Anxiety levels will be assessed using a Visual Analog Scale (VAS-A) during and after each session. If fail to achieve the desired anxiety score, participants will continue working with the study team until ready to progress. The final session includes in-person exposure to a real needle, aiming for voluntary vaccination or IV placement. Coping strategies will be discussed at the final session. Participants will be contacted for follow-up assessments at 6 and 12 weeks to evaluate long-term outcomes.

SUMMARY:
This case series study seeks to evaluate the use of a Spatial Computing Device and Augmented Reality (AR) and Virtual Reality (VR) as an exposure therapy modality for children and adolescents with needle and blood-injection-injury phobia. This study will take place at Lucile Packard Children's Hospital (LPCH) and Stanford Hospital (Stanford University, Palo Alto, CA).

DETAILED DESCRIPTION:
Needle phobia and Blood-Injection-Injury phobia are anxieties that are observed in children, adolescents, and adults undergoing medical/surgical procedures and the use of needles. These phobias can lead to an impediment of care for children or adolescents and may impact their ability to participate in care and/or receive essential treatments. This can lead to significant delays in treatment of individuals and medical trauma for patients who can only receive treatments/procedures using needles after undergoing sedation. Although treatment protocols exist for treating needle and blood-injection-injury phobia in adults, the literature regarding treatment in children and adolescents is limited. Additionally, the use of medications for management of needle phobia can lead to increased medical complications and may not resolve the underlying cause of needle phobia. Recent technological developments have led to the use of virtual reality exposure therapy (VRET) for treating needle and blood-injection-injury phobia, however few studies have been performed in children, and the literature regarding anxiety and clinical outcomes using this treatment modality is lacking in this population. Further, newly developed spatial computing and XR (Mixed Reality) devices have led to advancements in immersion and personalization of images/videos, and as such may lead to increased engagement and clinical efficacy for patients participating in VRET.

Here we propose to conduct a feasibility study to determine the safety and acceptability of using VRET for children and adolescents with needle and blood-injection-injury phobia undergoing procedures at LPCH and Stanford Hospital. This feasibility study will serve as the basis for a larger scale RCT to determine if VRET can serve as an alternative to traditional exposure therapy methods to improve anxiety related to these phobias, and increase engagement/participation with treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 8-17
2. Patients who complete a patient survey via QR code at Stanford blood draw and/or primary care clinics
3. Patients screened with the APA severity Measure for Specific Phobia (blood, needles, or injections), and have an individual phobia score rated as moderate, severe, or extreme (as described)

Exclusion Criteria:

1. Legal guardian not present to obtain consent
2. Adolescent with a significant neurological condition, or major developmental disability
3. Adolescent with active infection of the face or hand
4. A history of severe motion sickness
5. A history of seizures caused by flashing light
6. An impending surgery within the last 48 hours
7. Adolescents who wear glasses and cannot use contacts
8. Adolescents with myopia or astigmatism
9. Adolescents with physical disabilities that prevent them from using their hands
10. Patients with substance use disorder in past year
11. Patients screened with PHQ-9 and found to have a depression score greater than 15 and/or those with a score greater than 1 or above for questions related to suicidality
12. Patients screened with Child PTSD Symptom Scale Self-Report (CPSS-SR5) and found to have score greater than 31 (indicating likely PTSD diagnosis)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety symptoms related to needle phobia and BII | Baseline, immediately after the intervention, 6 and 12 weeks after completion of treatment
  APA severity Measure for Specific Phobia (APA-SMS) is a validated tool used to assess the severity of specific phobia symptoms, including needle and blood-injection-injury (BII) phobia. The scale has 10 items, rated on a 5-point Likert scale (0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme). The total score ranges from 0 - 40, with higher scores indicating greater severity of phobia. A change in symptom ratings from moderate/severe/extreme rating to mild/none indicates remission of symptoms by the end of intervention. The time to remission will be measured by the completion of sessions to reach remission, whether the participants complete the sessions as scheduled, or they need extra sessions.

SECONDARY OUTCOMES:
Skin Conductance Response Density (SCRD) | immediately before the first intervention, immediately after the last intervention
  Change in sympathetic response to a scripted discussion regarding use of a needle and needle being shown - administered at the beginning of the first session and at the end of the last session.
Parasympathetic response indexed by Respiratory sinus arrhythmia (RSA) | immediately before the first intervention, immediately after the last intervention
  Change in parasympathetic response to a scripted discussion regarding use of a needle and needle being shown. Measured via respiratory sinus arrhythmia (RSA) in hertz using chest biometric sensors in 30-second epochs.
Change in Anxiety after virtual exposure | Baseline, immediately after the intervention, up to 12-weeks
  Anxiety levels will be measured by a Visual Analogue Scale - Anxiety (VAS-A), where participants rate their anxiety in a scale ranging from 0-10, with 0 representing no anxiety to 10 representing extreme anxiety. Higher scores indicate higher anxiety levels.
Change in Anxiety after real exposure | during intervention, immediately after the intervention, up to 12-weeks
  Anxiety levels will be measured by a Visual Analogue Scale - Anxiety (VAS-A), where participants rate their anxiety in a scale ranging from 0-10, with 0 representing no anxiety to 10 representing extreme anxiety. Higher scores indicate higher anxiety levels.
User engagement | Immediately after final intervention
  User engagement will be measured by User Engagement Scale (UES) - Short. This scale consists of 12 items that participants will respond to, reflecting their feelings and interactions with the application or platform. Each item is rated on a Likert scale ranging from 1 to 5, where 1 indicates "strongly disagree" and 5 indicates "strongly agree."

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lulla, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Lucile Parkard Children's Hospital, Stanford, California, United States